CLINICAL TRIAL: NCT00060346
Title: Phase II Pilot Study Of Rituximab Plus CHOP In Patients With Newly Diagnosed Waldenstrom's Macroglobulinemia
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Newly Diagnosed Waldenstrom's Macroglobulinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000301634; U10CA021115 (NIH); E1A02 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; Rituximab; CHOP
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab + CHOP (Experimental): Rituximab 375 mg/m2 day 1 of a 21-day cycle, followed by:
  Cyclophosphamide 750 mg/m2 Doxorubicin 50 mg/m2 Vincristine 1.4 mg/m2 and Prednisone 100 mg/m2 daily
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Vincristine

INTERVENTIONS:
Biological: rituximab — Rituximab is given intravenously. The initial rate is 50 mg/hr for the 1st hour. If no toxicity, the rate may be escalated in 50 mg/hr increments at 30-minute intervals to a maximum of 400 mg/hr. If the first dose is well tolerated, the initial rate for subsequent dose is 100 mg/hr, increased in 100 mg/hr increments at 30-minute intervals, not to exceed 400 mg/hr. If the patient experiences fever and rigors, the antibody infusion is discontinued. The severity of the side effects should be evaluated. If the symptoms improve, the infusion is continued initially at half the previous rate. Following the antibody infusion, the intravenous line should be maintained for medications as needed. If there are no complications after one hour of observation, the intravenous line may be discontinued.
  Other Names: IDEC-C2B8; Chimeric anti-CD20 monoclonal antibody; Rituxan; NSC# 687451
Drug: cyclophosphamide — Cyclophosphamide will be given at a dosage of 750 mg/m² intravenously on day 1 of each cycle (1 cycle =21 days) for 6 cycles. Dose is based on surface area calculated based on actual body weight.
  The drug should be administered as a rapid IV infusion over 5 to 30 minutes.
  Other Names: Cytoxan; CTX; CPM; Neosar
Drug: Doxorubicin — Doxorubicin will be given intravenously at a dosage of 50 mg/m² on day 1 of each cycle for 6 cycles (1 cycle =21 days). Dose is based on surface area calculated based on actual body weight.
  Doxorubicin should be administered as a continuous infusion into tubing of a freely flowing intravenous line for 5 -15 minutes. Avoid extravasation.
  Other Names: Adriamycin; Rubex; Adriamycin RDF; Adriamycin PFS; hydroxydaunorubicin; ADR
Drug: Prednisone — Prednisone will be administered at 100 mg/m² orally, days 1-5 of each cycle for 6 cycles (1 cycle =21 days). Dose is based on surface area calculated based on actual body weight.
  Other Names: Deltasone; Orasone; Medicortone; Panasol-S; Liqui-Pred
Drug: Vincristine — Vincristine will be administered 1.4 mg/m² intravenously (Maximum dose = 2.0 mg) on day 1 of each cycle for 6 cycles (1 cycle =21 days). Dose is based on surface area calculated based on actual body weight.
  Given as IV push over 1 minute, using extravasation precautions.
  Other Names: Vinsacar PFS; vincristine sulfate; VCR; leucocristine; LCR

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining rituximab with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy works in treating patients with newly diagnosed Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with newly diagnosed Waldenstrom's macroglobulinemia treated with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone.
* Determine the associated toxic effects of this regimen, specifically the frequency of febrile neutropenia, in these patients.
* Determine the progression-free survival of patients treated with this regimen.
* Correlate baseline cytogenetic features and gene expression profiles with response in patients treated with this regimen.

OUTLINE: This is a pilot, multicenter study.

Patients receive rituximab intravenously (IV) over approximately 4 hours, cyclophosphamide IV over 5-30 minutes, doxorubicin IV over 5-15 minutes, and vincristine IV over 1 minute on day 1. Patients also receive oral prednisone on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ACTUAL ACCRUAL: A total of 16 patients were accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of Waldenstrom's macroglobulinemia confirmed by the presence of the following:

  * Bone marrow lymphoplasmacytosis with: > 10% lymphoplasmacytic cells OR aggregates or sheets of one of the following: lymphocytes, plasma cells or lymphoplasmacytic cells on the bone marrow biopsy (measured within 4 weeks prior to registration)
  * Measurable disease defined as a quantitative immunoglobulin M (IgM) monoclonal protein of > 1,000 mg/dL obtained within 4 weeks prior to registration
  * Cluster of differentiation 20 (CD20) positive stain of bone marrow or lymph node samples obtained < 8 weeks prior to registration
* Impaired bone marrow function due to infiltration by lymphoplasmacytic lymphoma, defined by 1 of the following:

  * Hemoglobin no greater than 11 g/dL
  * Serum viscosity level relative to water of at least 4.0 centipoise
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3
* Bilirubin no greater than 3.0 mg/dL
* Aspartate aminotransferase (AST) no greater than 3 times upper limit of normal
* Creatinine no greater than 3.0 mg/dL
* Age of 18 and over
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Must be symptomatic with 1 of the following:

  * Clinically significant anemia (hemoglobin no greater than 11 g/dL)
  * Bulky lymphadenopathy
  * Symptoms attributable to hyperviscosity (e.g., nose bleeding, gingival bleeding, or retinal hemorrhage)
* History of heart disease allowed only if 1 of the following is demonstrated by echocardiography, multigated acquisition scan (MUGA), exercise MUGA, or coronary catheterization:

  * Ejection fraction of at least 45%
  * Normal fractional shortening of the left ventricle
* Must have been tested for hepatitis B surface antigen within 2 weeks of registration
* Negative pregnancy test
* Fertile patients must use effective contraception

EXCLUSION CRITERIA:

* Prior treatment for Waldenstrom's macroglobulinemia
* Prior anti-CD20 therapy
* Concurrent steroids exceeding 10 mg prednisone (or equivalent) per day
* Prior irradiation if less than 4 weeks had elapsed prior to registration and the date of last treatment
* Prior anthracyclines
* Prior malignancy except curatively treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or other cancer curatively treated with surgery alone and from which patient has been disease free for at least 5 years
* Active heart disease
* Pregnant or nursing
* Myocardial infarction within the past 3 months
* Congestive heart failure
* Symptomatic ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-10-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafat Abonour, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (153):
- United States (153):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Abonour R, Zhang LA, Rajkumar V, et al.: Phase II pilot study of rituximab + CHOP in patients with newly diagnosed Waldenstroms macroglobulinemia, an Eastren Cooperative Oncology Group trial (study E1A02). [Abstract] Blood 110 (11): A-3616, 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on June 15, 2004, accrued its first patient on October 5, 2004, and closed due to slow accrual on April 26, 2007. Sixteen patients were accrued in this trial from Eastern Cooperative Oncology Group (ECOG) and Southwest Oncology Group (SWOG) institutions.
Period: Overall Study
Arm/Group | Rituximab + CHOP
Started | 16
Eligible and Treated | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab + CHOP
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 59.5 [44.1 to 78.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response to Treatment
Description: Objective response assessed using standard myeloma response criteria. Objective response is defined as a > 50% reduction in the quantitative IgM or M-Spike levels from baseline levels. Response must be documented by two measurements separated by at least 3 weeks.
Time Frame: Every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2-5 years from study entry, every 12 months if patient is 6-10 years from study entry
Population: All eligible and treated patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Rituximab + CHOP
Number analyzed (Participants) | 16
proportion of participants | 0.938 [0.736 to 0.997]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment.
Arm/Group | Rituximab + CHOP
Serious Adverse Events (participants affected / at risk) | 16/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + CHOP (N=16)
Allergic reaction (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Leukopenia (Investigations) | 8
Lymphopenia (Investigations) | 8
Neutropenia (Investigations) | 13
Cardiac-Left Ventricular Function (Cardiac disorders) | 1
Edema (General disorders) | 1
Hypotension (Vascular disorders) | 2
Thrombosis/Embolism (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Infection w/ Gr3-4 neutropenia (Infections and infestations) | 3
Infection w/o neutropenia (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Neuropathy-motor (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + CHOP (N=16)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 14
Leukopenia (Investigations) | 16
Lymphopenia (Investigations) | 15
Neutropenia (Investigations) | 15
Thrombocytopenia (Investigations) | 8
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Cardiac-Left Ventricular Function (Cardiac disorders) | 1
Edema (General disorders) | 3
Hypotension (Vascular disorders) | 2
Fatigue (General disorders) | 14
Fever (General disorders) | 2
Rigors/chills (General disorders) | 5
Sweating (Skin and subcutaneous tissue disorders) | 2
Weight gain (Investigations) | 1
Constitutional symptoms (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9
Bruising (Injury, poisoning and procedural complications) | 1
Flushing (Vascular disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Skin- Other (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 4
Taste disturbance (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2
Alkaline phosphatase increased (Investigations) | 2
Bilirubin increased (Investigations) | 1
SGOT increased (Investigations) | 5
Infection w/o neutropenia (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Dizziness/Lightheadedness (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 5
Anxiety/Agitation (Psychiatric disorders) | 2
Neuropathy-motor (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 11
Abdominal Pain (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Earache (Ear and labyrinth disorders) | 1
Headache (Nervous system disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain-other (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 4
Urinary Frequency/Urgency (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No